CLINICAL TRIAL: NCT01565460
Title: Bile and Bile Duct/Pancreatic Duct Brushings Database for Patients With Pancreato-biliary Stricture
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Mansour Parsi, MD, MD, The Cleveland Clinic
Other Study IDs: 11-976
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Pancreatic Duct Strictures; Biliary Duct Strictures
Keywords: pancreas; biliary; stricture
MeSH Terms: conditions — Constriction, Pathologic | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bile and bile duct/pancreatic duct brushings
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pancreatic/biliary strictures: Sample Collection: Patients with pancreatic/biliary stricture undergoing intervention will have samples of brushings and bile taken during the procedure.
  Interventions: Other: Sample Collection

INTERVENTIONS:
Other: Sample Collection — Sample Collection: bile and pancreatic duct brushings and fluid samples will be obtained from the pancreatic stricture during endoscopic retrograde cholangiopancreatic procedure.

SUMMARY:
The purpose of this study is to create a long-term storage of bile and brushings of pancreato-biliary duct in patients diagnosed with pancreato-biliary stricture for future research.

Recently, a lot of research has been done to test for certain markers in the bile and brushings to detect cancer in a stricture. The samples will be used to measure biomarkers (proteins) in biliary diseases.

DETAILED DESCRIPTION:
Recently, a lot of research has been done to test for certain markers like fluorescence in situ hybridization (FISH), digital image analysis (DIA), and quantifiable morphometric results in biliary stricture brushings. Recently, polysomy FISH has been studied as a promising marker in predicting cancer in a pancreato-biliary stricture. Many genetic, epigenetic, and protein alterations arise during pancreaticobiliary tumor process. The types of markers that have been commonly evaluated as diagnostic assays are mutations, chromosomal gains and losses, and DNA methylation alterations. However there are only a few studies in this area. Testing for these markers can help determine whether the narrowing or stricture in your bile duct is cancer or not.

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with pancreato-biliary stricture.
* Age >18 years
* Ability to provide an informed consent

Exclusion Criteria:

* Patients with altered mental status, who will not be able to provide an informed consent
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with pancreatic or biliary duct stricture who present for evaluation and intervention of their stricture
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Udayakumar Navaneethan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Navaneethan U, Parsi MA, Lourdusamy V, Bhatt A, Gutierrez NG, Grove D, Sanaka MR, Hammel JP, Stevens T, Vargo JJ, Dweik RA. Volatile organic compounds in bile for early diagnosis of cholangiocarcinoma in patients with primary sclerosing cholangitis: a pilot study. Gastrointest Endosc. 2015 Apr;81(4):943-9.e1. doi: 10.1016/j.gie.2014.09.041. Epub 2014 Dec 12. PMID 25500329
- [Derived] Navaneethan U, Parsi MA, Gutierrez NG, Bhatt A, Venkatesh PG, Lourdusamy D, Grove D, Hammel JP, Jang S, Sanaka MR, Stevens T, Vargo JJ, Dweik RA. Volatile organic compounds in bile can diagnose malignant biliary strictures in the setting of pancreatic cancer: a preliminary observation. Gastrointest Endosc. 2014 Dec;80(6):1038-45. doi: 10.1016/j.gie.2014.04.016. Epub 2014 Jun 11. PMID 24929484